CLINICAL TRIAL: NCT07086651
Title: Real-world Clinical Outcomes With Androgen Receptor Pathway Inhibitors (ARPIs) in Metastatic Castration-sensitive Prostate Cancer (mCSPC) in the Flatiron Health Electronic Health Records (EHR) Database
Brief Title: A Study to Learn About Two Medicines (Apalutamide and Enzalutamide) in People With Metastatic Castration-sensitive Prostate Cancer (mCSPC)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C3431053
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration Sensitive Prostate Cancer (mCSPC); Cancer of the Prostate; Prostate Neoplasms; Prostate Cancer
Keywords: enzalutamide; Xtandi; apalutamide; Erleada; mCSPC; metastatic castration-sensitive prostate cancer; treatment duration; metastatic hormone-sensitive prostate cancer; mHSPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; apalutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enzalutamide cohort: Patients initiating enzalutamide for mCSPC
  Interventions: Drug: Enzalutamide
- Apalutamide cohort: Patients initiating apalutamide for mCSPC
  Interventions: Drug: Apalutamide

INTERVENTIONS:
Drug: Enzalutamide — As provided in real-world setting
  Other Names: XTANDI
  Groups: Enzalutamide cohort
Drug: Apalutamide — As provided in real-world setting
  Other Names: ERLEADA
  Groups: Apalutamide cohort

SUMMARY:
The purpose of this study is to learn about how long apalutamide and enzalutamide are taken by men to treat mCSPC.

Prostate cancer is one of the most common cancers in men. The prostate is a gland in the male body that helps make semen. Metastatic cancer is a cancer that has spread to other parts of the body. Castration-sensitive prostate cancer means the cancer is being controlled by keeping the testosterone levels as low as would be expected if the testicles were removed by surgery.

This is a real-world study, not a clinical study. This means that researchers will look at what happens when men receive the treatments prescribed by their own doctor as part of their usual healthcare treatment. In this study, researchers will use information from cancer clinics (Flatiron Health electronic health records).

The study will include patients' information from the database for men who:

* Were identified to have mCSPC.
* Started treatment with apalutamide or enzalutamide (index date) for mCSPC.
* Were 18 years of age or older on the index date. Men in this study will be taking apalutamide or enzalutamide for treatment of their mCSPC. The study will compare how long men take apalutamide or enzalutamide. This study will use patient information from cancer clinics. Information from start of apalutamide or enzalutamide treatment until information is available in the database will be used to describe how long patients receive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male patients diagnosed with metastatic prostate cancer
* Initiated apalutamide or enzalutamide for the first-line treatment of metastatic castration-sensitive prostate cancer (mCSPC). Initiation date of first treatment defines the index date.
* Index date on or after 1 January 2020
* Evidence of androgen deprivation therapy (ADT) use between 90 days prior to the index date and 6 months following the index date
* Age ≥18 years on the index date -≥6 months of clinical activity following the index date, unless the patient died

Exclusion Criteria:

* Evidence of castration-resistance prior to the index date
* Received chemotherapy, androgen receptor pathway inhibitor, radiopharmaceuticals, immunotherapy, PARP inhibitor, or estrogens prior to the index date
* Evidence of ADT use between 1 year and 91 days prior to the index date
* Had a prior history of other cancers

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Men with metastatic castration-sensitive prostate cancer who initiated apalutamide or enzalutamide and met eligibility criteria will be included in the study. Patients will be identified from the Flatiron Health electronic health records database.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Treatment duration | Up to approximately 65 months
  Treatment duration will be defined as the time from index date to the discontinuation (i.e., addition of subsequent treatment, treatment gap of 90 days, death) of the index treatment for any reason. Patients without an event will be censored on the date of last confirmed clinical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3431053